CLINICAL TRIAL: NCT00737568
Title: A Phase 3b, Randomized, Double-Blind, Double-Dummy Study Evaluating the Antiviral Efficacy, Safety, and Tolerability of Tenofovir Disoproxil Fumarate (DF) Monotherapy Versus Emtricitabine Plus Tenofovir DF Fixed-Dose Combination Therapy in Subjects With Chronic Hepatitis B Who Are Resistant to Lamivudine
Brief Title: Tenofovir Disoproxil Fumarate (Tenofovir DF) Versus Emtricitabine/Tenofovir DF in Subjects Resistant to Lamivudine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-174-0121
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Results first posted 2013-04-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B
Keywords: Tenofovir DF; Emtricitabine; Chronic hepatitis B; Combination therapy
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir DF (Experimental): TDF plus placebo to match FTC/TDF
  Interventions: Drug: TDF; Drug: FTC/TDF Placebo
- FTC/TDF (Experimental): FTC/TDF plus placebo to match TDF
  Interventions: Drug: FTC/TDF; Drug: TDF Placebo

INTERVENTIONS:
Drug: TDF — Tenofovir disoproxil fumarate (tenofovir DF; TDF) 300 mg tablet administered orally once daily
  Other Names: Viread®
  Arms: Tenofovir DF
Drug: FTC/TDF — Emtricitabine (FTC)/TDF 200/300 mg fixed-dose combination tablet administered orally once daily
  Other Names: Truvada®
  Arms: FTC/TDF
Drug: TDF Placebo — TDF placebo tablet administered orally once daily
  Arms: FTC/TDF
Drug: FTC/TDF Placebo — FTC/TDF placebo tablet administered orally once daily
  Arms: Tenofovir DF

SUMMARY:
The aim of therapy for the treatment of chronic hepatitis B virus (HBV) is to maintain suppression of viral replication to prevent the emergence of complications, which requires long-term therapy. Durable suppression of viral replication is achieved in the treatment of chronic viral diseases by preventing of the emergence of drug-resistant mutations. The clinical guidelines for the management of lamivudine resistant patients are variable. Some recommend switching to another agent without cross-resistance, while others recommend adding on another agent without cross-resistance. Limited clinical data exists to demonstrate whether tenofovir disoproxil fumarate (tenofovir DF; TDF) is an effective monotherapy for lamivudine resistant patients or if it should be used as part of a combination therapy regimen.

This study is designed to evaluate the effectiveness, safety, and tolerability of tenofovir DF monotherapy versus emtricitabine (FTC)/tenofovir DF combination therapy in participants with chronic HBV with lamivudine resistance (presence of the rtM204I/V mutation with or without the rtL180M mutation) over a 240-week period. Participants in this study must be receiving lamivudine treatment at the time of enrollment.

ELIGIBILITY:
Inclusion Criteria

* Chronic HBV infection, defined as positive serum HBsAg for at least 6 months
* 18 through 75 years of age, inclusive
* HBV DNA ≥ 10^3 IU/mL
* Receiving treatment with lamivudine with confirmation of HBV reverse transcriptase mutation(s) known to confer resistance to lamivudine (rtM204I/V with or without rtL180M) by central laboratory assessment prior to randomization; adefovir dipivoxil treatment of ≤ 48 weeks at the time of screening (inclusive of combination adefovir dipivoxil + lamivudine at entry) was allowed
* Willing and able to provide written informed consent
* Negative serum pregnancy test (for females of childbearing potential only)
* Calculated creatinine clearance ≥ 50 mL/min
* Hemoglobin ≥ 10 g/dL
* Neutrophils ≥ 1000 /mm^3
* No prior oral HBV therapy with approved nucleotide and/or nucleoside therapy or other investigational agents for HBV infection other than lamivudine or adefovir dipivoxil

Exclusion Criteria

* Pregnant women, women who are breast feeding or who believe they may wish to become pregnant during the course of the study
* Males and females of reproductive potential who are not willing to use an effective method of contraception during the study
* Alanine aminotransferase (ALT) ≥ 10 × the upper limit of the normal range (ULN)
* Decompensated liver disease
* Interferon or pegylated interferon therapy within 6 months of the screening visit
* Alpha fetoprotein > 50 ng/mL
* Evidence of hepatocellular carcinoma
* Coinfection with hepatitis C virus, HIV, or hepatitis D virus
* Significant renal, cardiovascular, pulmonary, or neurological disease
* Received solid organ or bone marrow transplantation
* Receiving therapy with immunomodulators (eg, corticosteroids, etc.), investigational agents, nephrotoxic agents, or agents susceptible of modifying renal excretion
* Proximal tubulopathy
* Known hypersensitivity to the study drugs, the metabolites or formulation excipients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, PharmD, Study Director — Gilead Sciences
Locations (56):
- United States (3):
  - Bradenton, Florida
  - Flushing, New York
  - Philadelphia, Pennsylvania
- Austria (2):
  - Innsbruck
  - Vienna
- Bulgaria (2):
  - Sofia
  - Varna
- Canada (3):
  - Vancouver, British Columbia
  - Winnepeg, Manitoba
  - Toronto, Ontario
- Czechia (4):
  - Brno
  - Pilsen
  - Prague
  - Ústí nad Labem
- Germany (8):
  - Ulm, Baden-Wurttemberg
  - Berlin
  - Düsseldorf
  - Essen
  - Frankfurt
  - Hamburg
  - Hanover
  - Stuttgart
- Greece (3):
  - Larissa
  - Pátrai
  - Thessaloniki
- Hungary (4):
  - Budapest
  - Debrecen
  - Gyula
  - Kasposvar
- New Zealand (3):
  - Auckland
  - Hamilton
  - Wellington
- Poland (8):
  - Bialystok
  - Bydgoszcz
  - Chorzów
  - Krakow
  - Lodz
  - Szczecin
  - Warsaw
  - Wroclaw
- Romania (5):
  - Lasi, Judetul Lasi
  - Timișoara, Timiș County
  - Bucharest
  - Cluj-Napoca
  - Constanța
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Sad
- Seville, Spain
- Turkey (Türkiye) (6):
  - Ankara
  - Bursa
  - Izmir
  - Samsun
  - Trabzon
  - Üsküdar

REFERENCES:
- [Result] Corsa AC, Liu Y, Flaherty JF, Mitchell B, Fung SK, Gane E, Miller MD, Kitrinos KM. No resistance to tenofovir disoproxil fumarate through 96 weeks of treatment in patients with lamivudine-resistant chronic hepatitis B. Clin Gastroenterol Hepatol. 2014 Dec;12(12):2106-12.e1. doi: 10.1016/j.cgh.2014.05.024. Epub 2014 Jun 11. PMID 24929235
- [Result] Liu Y, Fung S, Gane EJ, Dinh P, Flaherty JF, Svarovskaia ES, Miller MD, Kitrinos KM. Evaluation of HBV DNA decay kinetics in patients containing both rtM204V/I mutant and wild-type HBV subpopulations during tenofovir DF (TDF) monotherapy or combination therapy with emtricitabine (FTC)/TDF. J Med Virol. 2014 Sep;86(9):1473-81. doi: 10.1002/jmv.23982. Epub 2014 May 23. PMID 24861361
- [Result] Fung S, Kwan P, Fabri M, Horban A, Pelemis M, Hann HW, Gurel S, Caruntu FA, Flaherty JF, Massetto B, Dinh P, Corsa A, Subramanian GM, McHutchison JG, Husa P, Gane E. Randomized comparison of tenofovir disoproxil fumarate vs emtricitabine and tenofovir disoproxil fumarate in patients with lamivudine-resistant chronic hepatitis B. Gastroenterology. 2014 Apr;146(4):980-8. doi: 10.1053/j.gastro.2013.12.028. Epub 2013 Dec 22. PMID 24368224
- [Derived] Fung S, Kwan P, Fabri M, Horban A, Pelemis M, Hann HW, Gurel S, Caruntu FA, Flaherty JF, Massetto B, Kim K, Kitrinos KM, Subramanian GM, McHutchison JG, Yee LJ, Elkhashab M, Berg T, Sporea I, Yurdaydin C, Husa P, Jablkowski MS, Gane E. Tenofovir disoproxil fumarate (TDF) vs. emtricitabine (FTC)/TDF in lamivudine resistant hepatitis B: A 5-year randomised study. J Hepatol. 2017 Jan;66(1):11-18. doi: 10.1016/j.jhep.2016.08.008. Epub 2016 Aug 18. PMID 27545497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and New Zealand. The first participant was screened on 30 September 2008. The last study visit occurred on 09 February 2015.
Pre-assignment Details: 752 participants were screened. Randomization was stratified by hepatitis B e antigen (HBeAg) status (negative or positive) and alanine aminotransferase (ALT) level (≥ 2 × upper limit of normal [ULN] or < 2 × ULN) at screening.
Groups:
- Tenofovir DF: Tenofovir disoproxil fumarate (tenofovir DF; TDF) 300 mg tablet once daily plus emtricitabine (FTC)/TDF placebo tablet once daily
- FTC/Tenofovir DF: FTC/TDF 200/300 mg tablet once daily plus TDF placebo tablet once daily
Period: Treatment Period Through Week 240
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Started | 141 | 139
Completed | 121 | 118
Not Completed | 20 | 21
Not completed — Investigator's Discretion | 6 | 5
Not completed — Withdrew Consent | 5 | 6
Not completed — Safety, Tolerability, or Efficacy Reason | 3 | 4
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 2 | 3
Not completed — Study Discontinued by Sponsor | 1 | 0
Period: Treatment-Free Follow-up (TFFU) Period
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Started | 38 (1 participant not completing the 240 week treatment period enrolled in the TFFU period.) | 37 (4 participants not completing the 240 week treatment period enrolled in the TFFU period.)
Completed | 12 | 19
Not Completed | 26 | 18
Not completed — Started Commercial Therapy | 25 | 17
Not completed — Death | 0 | 1
Not completed — Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tenofovir DF: TDF 300 mg tablet once daily plus FTC/TDF placebo tablet once daily
- Total: Total of all reporting groups
Arm/Group | Tenofovir DF | FTC/Tenofovir DF | Total
Number analyzed (Participants) | 141 | 139 | 280
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (13.63) | 46.3 (13.56) | 46.7 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 69
  Male | 104 | 107 | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 138 | 137 | 275
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 52 | 42 | 94
  Black or African American | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  White | 83 | 89 | 172
  Other | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  Austria | 2 | 3 | 5
  Bulgaria | 2 | 5 | 7
  Canada | 47 | 43 | 90
  Czech Republic | 9 | 7 | 16
  Germany | 2 | 0 | 2
  Greece | 2 | 1 | 3
  Hungary | 4 | 3 | 7
  New Zealand | 7 | 10 | 17
  Poland | 13 | 19 | 32
  Romania | 17 | 14 | 31
  Serbia | 17 | 19 | 36
  Spain | 1 | 1 | 2
  Turkey | 15 | 13 | 28
  United States | 3 | 1 | 4
ALT Normal at Baseline [Number; unit: participants] — The ULN was 43 U/L for males and 34 U/L for females aged 18 to < 69, and 35 U/L for males and 32 U/L for females aged ≥ 69.
  participants
    Abnormal | 79 | 83 | 162
    Normal | 62 | 56 | 118
Hepatitis B Virus (HBV) DNA Level at Baseline [Mean (Standard Deviation); unit: log_10 copies/mL] | 6.40 (1.826) | 6.53 (1.968) | 6.46 (1.896)
HBV e Antigen (HBeAg) Status at Baseline [Number; unit: participants]
  Negative | 76 | 71 | 147
  Positive | 65 | 68 | 133

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Week 96
Time Frame: Week 96
Population: Full Analysis Set: participants were randomized and received at least 1 dose of study drug. The missing = failure method was used in which participants with missing data were considered to have failed to achieve the endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
percentage of participants | 89.4 | 86.3
Statistical Analysis 1: Comparison: Tenofovir DF vs FTC/Tenofovir DF; The null hypothesis is that there is no difference between the FTC/TDF and TDF treatment groups. The alternative hypothesis is that there is a difference between the FTC/TDF and TDF treatment groups. These hypotheses were evaluated using a Cochran-Mantel-Haenszel (CMH) test, controlling for randomization strata, with the missing = failure method in which participants with missing data were considered to have failed to achieve the endpoint; Test type: Superiority or Other; p = 0.43, Cochran-Mantel-Haenszel — The p-value for the two-sided Cochran-Mantel-Haenszel test was controlled for strata (HBeAg status and ALT level)

2. Secondary Outcome: Percentage of Participants With HBV DNA < 400 Copies/mL at Weeks 48, 144, 192, and 240
Time Frame: Weeks 48, 144, 192, and 240
Population: Full Analysis Set, missing = failure method
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
percentage of participants
  Week 48 | 81.6 | 84.2
  Week 144 | 87.2 | 84.9
  Week 192 | 86.5 | 85.6
  Week 240 | 83.0 | 82.7

3. Secondary Outcome: Percentage of Participants With HBV DNA < 169 Copies/mL at Weeks 48, 96, 144, 192, and 240
Time Frame: Weeks 48, 96, 144, 192, and 240
Population: Full Analysis Set, missing = failure method
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
percentage of participants
  Week 48 | 76.6 | 77.7
  Week 96 | 85.8 | 83.5
  Week 144 | 86.5 | 84.9
  Week 192 | 85.1 | 84.2
  Week 240 | 81.6 | 82.0

4. Secondary Outcome: HBV DNA Level at Weeks 48, 96, 144, 192, and 240
Time Frame: Weeks 48, 96, 144, 192, and 240
Population: Full analysis set; participants with HBV DNA measurements at the given time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
log10 copies/mL
  Week 48 (TDF: n=130; FTC/TDF: n=133) | 2.42 (0.542) | 2.48 (0.887)
  Week 96 (TDF: n=132; FTC/TDF: n=127) | 2.29 (0.254) | 2.28 (0.241)
  Week 144 (TDF: n=128; FTC/TDF: n=123) | 2.26 (0.173) | 2.29 (0.541)
  Week 192 (TDF: n=126; FTC/TDF: n=119) | 2.25 (0.135) | 2.23 (0.027)
  Week 240 (TDF: n=118; FTC/TDF: n=116) | 2.23 (0.052) | 2.26 (0.376)

5. Secondary Outcome: Percentage of Participants With Normal ALT at Weeks 48, 96, 144, 192, and 240
Description: Normal ALT was defined as having a value less than or equal to the ULN. The ULN was 43 U/L for males and 34 U/L for females aged 18 to < 69, and 35 U/L for males and 32 U/L for females aged ≥ 69.
Time Frame: Weeks 48, 96, 144, 192, and 240
Population: Full Analysis Set, missing = failure method
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
percentage of participants
  Week 48 | 67.4 | 69.8
  Week 96 | 70.2 | 69.8
  Week 144 | 70.2 | 75.5
  Week 192 | 75.9 | 76.3
  Week 240 | 71.6 | 71.9

6. Secondary Outcome: Percentage of Participants With HBeAg Loss at Weeks 48, 96, 144, 192, and 240
Description: The percentage of participants who were HBeAg positive at baseline and who had HBeAg Loss at the given time point was summarized. Loss of HBeAg was defined as change of detectable HBeAg from positive to negative.
Time Frame: Baseline; Weeks 48, 96, 144, 192, and 240
Population: Participants in the Full Analysis Set who were HBeAg positive at baseline were analyzed using the missing = failure method.
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 65 | 68
percentage of participants
  Week 48 | 9.2 | 5.9
  Week 96 | 15.4 | 13.2
  Week 144 | 23.1 | 17.6
  Week 192 | 21.5 | 14.7
  Week 240 | 24.6 | 19.1

7. Secondary Outcome: Percentage of Participants With Seroconversion to Antibody Against HBeAg (Anti-HBe) at Weeks 48, 96, 144, 192, and 240
Description: The percentage of participants who were HBeAg positive at baseline and who had seroconversion to anti-HBe at the given time point was summarized. Seroconversion to anti-HBe was defined as change of detectable antibody to HBeAg from negative to positive.
Time Frame: Baseline; Weeks 48, 96, 144, 192, and 240
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 65 | 68
percentage of participants
  Week 48 | 6.2 | 4.4
  Week 96 | 10.8 | 10.3
  Week 144 | 12.3 | 11.8
  Week 192 | 10.8 | 10.3
  Week 240 | 12.3 | 10.3

8. Secondary Outcome: Percentage of Participants With HBV Surface Antigen (HBsAg) Loss at Weeks 48, 96, 144, 192, and 240
Description: The percentage of participants with HBsAg Loss at the given time point was summarized. Loss of HBsAg was defined as change of detectable HBsAg from positive to negative.
Time Frame: Baseline; Weeks 48, 96, 144, 192, and 240
Population: Full Analysis Set, missing = failure method
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
percentage of participants
  Week 48 | 0.0 | 0.7
  Week 96 | 0.0 | 0.7
  Week 144 | 0.7 | 1.4
  Week 192 | 0.7 | 2.9
  Week 240 | 1.4 | 2.9

9. Secondary Outcome: Percentage of Participants With Seroconversion to Antibody Against HBV Surface Antigen (Anti-HBs) at Weeks 48, 96, 144, 192, and 240
Description: The percentage of participants with seroconversion to anti-HBs at the given time point was summarized. Seroconversion to anti-HBs was defined as change of detectable antibody to HBsAg from negative to positive.
Time Frame: Baseline; Weeks 48, 96, 144, 192, and 240
Population: Full Analysis Set, missing = failure method
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
percentage of participants
  Week 48 | 0.0 | 0.0
  Week 96 | 0.0 | 0.0
  Week 144 | 0.0 | 0.7
  Week 192 | 0.0 | 0.7
  Week 240 | 0.0 | 0.7

10. Secondary Outcome: Percentage of Participants With Virologic Breakthrough at Weeks 48, 96, 144, 192, and 240
Description: The percentage of participants with virologic breakthrough at the given time point was summarized. Virologic breakthrough was defined as having two consecutive 1.0 log10 or greater increases in serum HBV DNA from on-treatment nadir, or two consecutive HBV DNA values ≥ 400 copies/mL after being < 400 copies/mL.
Time Frame: Baseline; Weeks 48, 96, 144, 192, and 240
Population: Full Analysis Set; the missing-equals-excluded method was used in which participants with missing data were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
percentage of participants
  Week 48 (TDF: n=130; FTC/TDF: n=133) | 0.0 | 0.8
  Week 96 (TDF: n=132; FTC/TDF: n=127) | 0.0 | 0.0
  Week 144 (TDF: n=128; FTC/TDF: n=123) | 0.8 | 0.8
  Week 192 (TDF: n=126; FTC/TDF: n=119) | 0.8 | 0.0
  Week 240 (TDF: n=118; FTC/TDF: n=116) | 0.0 | 0.0

11. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD) of the Spine at Weeks 24, 48, 72, 96, 144, 192, and 240
Description: BMD is calculated as grams per cubic centimeter (g/cm^2); the mean (SD) percentage change is presented.
Time Frame: Baseline; Weeks 24, 48, 72, 96, 144, 192, and 240
Population: Participants in the Safety Analysis Set (randomized and received at least 1 dose of study drug) with spine BMD measurements at the given time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
percentage change
  % Change at Week 24 (TDF: n=132; FTC/TDF: n=127) | -1.74 (2.867) | -1.83 (2.565)
  % Change at Week 48 (TDF: n=126; FTC/TDF: n=121) | -1.68 (3.094) | -1.73 (2.944)
  % Change at Week 72 (TDF: n=123; FTC/TDF: n=119) | -1.35 (3.337) | -1.95 (2.977)
  % Change at Week 96 (TDF: n=126; FTC/TDF: n=114) | -1.24 (3.761) | -1.72 (3.269)
  % Change at Week 144 (TDF: n=123; FTC/TDF: n=110) | -1.36 (3.810) | -1.63 (3.591)
  % Change at Week 192 (TDF: n=120; FTC/TDF: n=106) | -1.32 (4.237) | -1.60 (4.628)
  % Change at Week 240 (TDF: n=115; FTC/TDF: n=102) | -0.83 (4.490) | -1.15 (5.130)

12. Secondary Outcome: Percent Change From Baseline in BMD of the Hip at Weeks 24, 48, 72, 96, 144, 192, and 240
Description: BMD is calculated as g/cm^2; the mean (SD) percentage change is presented.
Time Frame: Baseline; Weeks 24, 48, 72, 96, 144, 192, and 240
Population: Participants in the Safety Analysis Set with hip BMD measurements at the given time point were included in the analysis.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
percentage change
  % Change at Week 24 (TDF: n=130; FTC/TDF: n=127) | -0.71 (1.724) | -0.59 (1.835)
  % Change at Week 48 (TDF: n=126; FTC/TDF: n=118) | -1.15 (2.120) | -1.00 (2.063)
  % Change at Week 72 (TDF: n=121; FTC/TDF: n=115) | -1.59 (2.507) | -1.61 (2.525)
  % Change at Week 96 (TDF: n=125; FTC/TDF: n=112) | -1.70 (2.617) | -1.77 (2.801)
  % Change at Week 144 (TDF: n=120; FTC/TDF: n=107) | -2.02 (3.030) | -1.91 (3.281)
  % Change at Week 192 (TDF: n=116; FTC/TDF: n=105) | -2.33 (3.190) | -2.41 (3.783)
  % Change at Week 240 (TDF: n=111; FTC/TDF: n=100) | -2.46 (3.191) | -2.63 (3.872)

13. Secondary Outcome: Development of Drug-resistant Mutations (DRMs)
Description: The development of DRMs was summarized, either as development of new DRMs or enrichment of existing DRMs.
Time Frame: Baseline to Week 240
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Number analyzed (Participants) | 141 | 139
participants
  New tenofovir DF DRMs | 0 | 0
  Enrichment of tenofovir DF DRMs | 0 | 0
  New FTC DRMs | 0 | 0
  Enrichment of FTC DRMs | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline through end of study drug treatment (average exposure 220 weeks) plus 30 days
Description: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug.
Arm/Group | Tenofovir DF | FTC/Tenofovir DF
Serious Adverse Events (participants affected / at risk) | 23/141 | 21/139
Other Adverse Events (participants affected / at risk) | 109/141 | 105/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF (N=141) | FTC/Tenofovir DF (N=139)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bone tuberculosis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF (N=141) | FTC/Tenofovir DF (N=139)
Abdominal pain (Gastrointestinal disorders) | 6 | 7
Abdominal pain upper (Gastrointestinal disorders) | 8 | 12
Diarrhoea (Gastrointestinal disorders) | 13 | 7
Nausea (Gastrointestinal disorders) | 12 | 11
Fatigue (General disorders) | 14 | 15
Pyrexia (General disorders) | 8 | 5
Seasonal allergy (Immune system disorders) | 8 | 3
Influenza (Infections and infestations) | 14 | 10
Nasopharyngitis (Infections and infestations) | 24 | 20
Creatinine renal clearance decreased (Investigations) | 2 | 7
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 15
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 8
Dizziness (Nervous system disorders) | 7 | 8
Headache (Nervous system disorders) | 23 | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Hypertension (Vascular disorders) | 7 | 9

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years